CLINICAL TRIAL: NCT01716637
Title: Open Label,Crossover,Pilot Study to Assess the Efficacy & Safety of Perispinal Admin.of Etanercept(Enbrel®) in Comb.w/Nutritional Supplements vs. Nutritional Supplements Alone in Subj. w/Mild to Mod. Alzheimer's Disease Receiving Std. Care.
Brief Title: Short Term Efficacy and Safety of Perispinal Administration of Etanercept in Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Life Extension Foundation Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: CL025
Record Dates: First submitted 2012-10-05; First posted 2012-10-30 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Dementia; Cognitive decline; Cognitive disorder; Degenerative brain disease; Cognitive impairment; Memory loss; TNF-alpha
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction; Memory Disorders | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Etanercept (Active Comparator): 25 mg administered weekly for 6 weeks
  Interventions: Biological: Etanercept; Dietary Supplement: Curcum.Luteol.Theaflav.Lip.Acid,FishOil,Quercet.,Resveratr.
- Nutritional Supplements (Active Comparator): Nutritional supplements administered daily for 6 weeks in each period as well as an additional 12 weeks following visit 15.
  Interventions: Dietary Supplement: Curcum.Luteol.Theaflav.Lip.Acid,FishOil,Quercet.,Resveratr.

INTERVENTIONS:
Biological: Etanercept
  Other Names: Enbrel®
  Arms: Etanercept
Dietary Supplement: Curcum.Luteol.Theaflav.Lip.Acid,FishOil,Quercet.,Resveratr.
  Other Names: Super Bio-Curcumin; Super Omega-3; Optimized Quercetin; Optimized Resveratrol

SUMMARY:
While the cause of AD is still unknown, evidence suggests it develops because of a complex series of events in the brain that occur over time. Two pathways possibly involved in development of AD are inflammation and oxidative stress. Scientists have linked chronic inflammatory events in the brain with the onset and progression of Alzheimer's Disease. Oxidative stress has also been implicated in the pathogenesis of a number of neurological disorders including Alzheimer's Disease.

Etanercept (Enbrel®) is an approved drug for the treatment of several forms of arthritis when administered by injection. Some research suggests that etanercept, when administered by injection into the tissues close to the spinal column (perispinally), may modulate certain aspects of the immune system and provide some beneficial effect for people with Alzheimer's disease. Studies suggest that supplementation with specific nutrients may also have a positive effect in support of cognitive function.

This study will be conducted at one research office with volunteers who have been diagnosed with mild to moderate Alzheimer's disease. Each qualifying participant will be randomly assigned to receive an etanercept injection plus nutritional supplements for 6 weeks followed by a crossover and a washout period of 4 weeks to then receiving nutritional supplements alone or vice versa for another 6 weeks.

Participants will undergo blood and urine safety assessments at the beginning and end of each 6 week treatment period. During 4 of the 6 weekly visits in the treatment period with the injections, you will complete the cognitive tests twice; once before and once 2 hours after the injection. During 4 of the 6 weekly visits in the treatment period without the injections, you will also complete the cognitive tests twice; once before and once 2 hours after being asked to lie down onto a table for 5 minutes. You will be allowed to continue your standard of care for Alzheimer's disease throughout your participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject is aged 60-85 years
* Subject has a diagnosis of Alzheimer's disease according to the NINCDS- ADRDA criteria (National Institute of Neurological and Communicative Disorders and Stroke NINCDS] and Alzheimer's Disease and Related Disorders Association [ADRDA]).
* Subject is not institutionalized (for example, lives independently, lives independently in a residential home for the elderly, or is a day patient at a care center)
* Subject has a Hachinski Ischemia Score of ≤ 4.
* Subject has a total MoCA score of < 26 at screening.
* Subject has an MMSE score of 11 to 24 at screening.
* Subject has an ADAS-cog score of 12 to 25 at screening.
* Subject has experienced a gradual and progressive cognitive decline in the 6 months before the screening visit.
* Subject provides informed consent to participate in the study or has a legally acceptable representative who provides consent.
* Subject has a responsible caregiver who consents to supporting the subject in his/her study participation (for example, by accompanying the subject on each study visit).
* Subject is surgically sterile, agrees to use an acceptable method of birth control as defined in section 5.4 or, for females, is post- menopausal.
* Subject agrees to stop taking any vitamin, mineral, or dietary supplements he/she is currently taking that have any components of the nutritional supplements utilized in the study at least 7 days before randomization (Visit 2) and agrees to not use any new vitamin, mineral, or dietary supplement product other than those provided by the investigator until after the subject is discharged from the study.

Exclusion Criteria:

* A neurologic disorder, such as seizures, multiple sclerosis, neurodegenerative disorders (eg, Parkinson's disease), or dementia other than Alzheimer's type (including that caused by small strokes or cerebrovascular disease)
* Cognitive impairment from any condition other than Alzheimer's disease, such as that resulting from acute cerebral trauma, cerebral damage due to a lack of oxygen, infections such as meningitis or AIDS, significant endocrine or metabolic disease, mental retardation, or a brain tumor
* Cardiovascular or cerebrovascular disease, such as congestive heart failure, uncontrolled hypertension (BP ≥ 140/90 mmHg at screening), and a history of stroke
* Renal impairment/disease, defined as serum creatinine > 1.5 mg/dL
* Hepatic impairment, defined as Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) > 3 times the upper limit of normal OR has a history of a positive blood screen for hepatitis B surface antigen or hepatitis C antibody.
* Type I or II diabetes mellitus
* Significant or uncontrolled psychiatric disease
* Gastrointestinal disease, such as active peptic ulcer, gallstones, gallbladder disease, or biliary tract obstruction, or a history of cholecystectomy
* Hematologic disorders
* Pulmonary or lung disorders
* Immune system disorder, such as HIV/AIDS
* History of cancer within 10 years before screening (except localized skin cancer without metastases or in situ cervical cancer)
* History of chronic or recurrent infection (including tuberculosis) OR, in the 7 days before Visit 2 (randomization), any known infection or body temperature > 38.6º C (101.5º F)
* Subject is pregnant or breastfeeding at screening.
* Subject has intolerance or allergy to Enbrel®, latex, or any of Enbrel's components.
* Subject is currently consuming more than 6 standard alcoholic beverages a week. A standard alcoholic beverage is defined as 12 ounces of beer, 5 ounces of wine, or 1.5 ounces of liquor.
* Subject is currently taking and unable or unwilling to stop taking anticoagulant or antiplatelet herbs and supplements such as angelica, clove, danshen, garlic, ginger, ginkgo, Panax ginseng, red clover, or willow for at least 7 days before the randomization visit (Visit 2) and throughout the study.
* Subject is currently taking and unable or unwilling to stop taking any of the prohibited medications in protocol section 5.3.2 for at least 7 days before the randomization visit (Visit 2) and throughout the study.
* Subject had major surgery within the 4 weeks before screening.
* Subject has any condition or abnormality that, in the opinion of the investigator, would compromise the safety of the subject or the quality of the study data.
* Subject is participating or has participated in another research study within 30 days before the screening visit
* Subject or subject's caregiver is unable or unwilling to comply with the study procedures.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2010-02; Primary Completion 2015-10 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Difference in effects of treatment for 6 weeks with etanercept + nutritional supplements versus nutritional supplements alone on the Mini-Mental Status Examination (MMSE) score. | 16 weeks

SECONDARY OUTCOMES:
Difference in the effects of treatment for 6 weeks with etanercept + nutritional supplements versus nutritional supplements alone on the Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-cog) score. | 16 weeks
Difference in the effects of treatment for 6 weeks with etanercept + nutritional supplements versus nutritional supplements alone on the Montreal Cognitive Assessment (MoCA) score. | 16 weeks

OTHER OUTCOMES:
Difference in the effects of treatment for 6 weeks as well as an additional 12 weeks following visit 15 with nutritional supplementation alone on the MMSE score. | 28 weeks
Difference in short term effects of etanercept on the MMSE score before and two hours after perispinal administration of etanercept. | 16 weeks
To determine the safety and tolerability of nutritional supplements with perispinal adminstration of etanercept, as measured by various laboratory markers, vital signs (blood pressure and heart rate), and adverse events. | 16 weeks
Difference in the effects of treatment for 6 weeks as well as an additional 12 weeks following visit 15 with nutritional supplementation alone on the ADAS-cog score. | 28 weeks
Difference in the effects of treatment for 6 weeks as well as an additional 12 weeks following visit 15 with nutritional supplementation alone on the MoCA score. | 28 weeks
Difference in short term effects of etanercept on the ADAS-cog score before and two hours after perispinal administration of etanercept. | 16 weeks
Difference in short term effects of etanercept on the MoCA score before and two hours after perispinal administration of etanercept. | 16 weeks
To determine the safety and tolerability of nutritional supplements without perispinal adminstration of etanercept, as measured by various laboratory markers, vital signs (blood pressure and heart rate), and adverse events. | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul H. Wand, M.D., Principal Investigator — Paul H. Wand M.D., P.A.; Mark L. Brody, M.D., Principal Investigator — Brain Matters Research Inc.
Locations (2):
- United States (2):
  - Paul H. Wand M.D., P.A., Coral Springs, Florida
  - Brain Matters Research, Delray Beach, Florida

REFERENCES:
- [Background] Centers for Disease Control and Prevention website. CDC Features: Alzheimer's Disease. http://www.cdc.gov/Features/Alzheimers/. 12-15-2008. 6-23-2009.
- [Background] Mrak RE, Griffin WS. Interleukin-1, neuroinflammation, and Alzheimer's disease. Neurobiol Aging. 2001 Nov-Dec;22(6):903-8. doi: 10.1016/s0197-4580(01)00287-1. PMID 11754997
- [Background] Alzheimer's Disease Education & Referral (ADEAR) Center, National Institutes of Health. Alzheimer's Disease Fact Sheet. 2008.
- [Background] Mrak RE, Griffin WS. Glia and their cytokines in progression of neurodegeneration. Neurobiol Aging. 2005 Mar;26(3):349-54. doi: 10.1016/j.neurobiolaging.2004.05.010. PMID 15639313
- [Background] Tarkowski E, Andreasen N, Tarkowski A, Blennow K. Intrathecal inflammation precedes development of Alzheimer's disease. J Neurol Neurosurg Psychiatry. 2003 Sep;74(9):1200-5. doi: 10.1136/jnnp.74.9.1200. PMID 12933918
- [Background] McGeer PL, McGeer EG. Local neuroinflammation and the progression of Alzheimer's disease. J Neurovirol. 2002 Dec;8(6):529-38. doi: 10.1080/13550280290100969. PMID 12476347
- [Background] Kaur C, Ling EA. Antioxidants and neuroprotection in the adult and developing central nervous system. Curr Med Chem. 2008;15(29):3068-80. doi: 10.2174/092986708786848640. PMID 19075654
- [Background] Tobinick E, Gross H, Weinberger A, Cohen H. TNF-alpha modulation for treatment of Alzheimer's disease: a 6-month pilot study. MedGenMed. 2006 Apr 26;8(2):25. PMID 16926764
- [Background] Tarkowski E, Liljeroth AM, Minthon L, Tarkowski A, Wallin A, Blennow K. Cerebral pattern of pro- and anti-inflammatory cytokines in dementias. Brain Res Bull. 2003 Aug 15;61(3):255-60. doi: 10.1016/s0361-9230(03)00088-1. PMID 12909295
- [Background] Laws SM, Perneczky R, Wagenpfeil S, Muller U, Forstl H, Martins RN, Kurz A, Riemenschneider M. TNF polymorphisms in Alzheimer disease and functional implications on CSF beta-amyloid levels. Hum Mutat. 2005 Jul;26(1):29-35. doi: 10.1002/humu.20180. PMID 15895461
- [Background] Tobinick EL, Gross H. Rapid improvement in verbal fluency and aphasia following perispinal etanercept in Alzheimer's disease. BMC Neurol. 2008 Jul 21;8:27. doi: 10.1186/1471-2377-8-27. PMID 18644112
- [Background] Becker RE. Modifying clinical trial designs to test treatments for clinical significance in individual patients. Clin Drug Invest 2001:21:727-733.
- [Background] Griffin WS. Perispinal etanercept: potential as an Alzheimer therapeutic. J Neuroinflammation. 2008 Jan 10;5:3. doi: 10.1186/1742-2094-5-3. PMID 18186919
- [Background] Tobinick E. Perispinal etanercept for neuroinflammatory disorders. Drug Discov Today. 2009 Feb;14(3-4):168-77. doi: 10.1016/j.drudis.2008.10.005. Epub 2008 Dec 6. PMID 19027875
- [Background] Tobinick E. Perispinal etanercept for treatment of Alzheimer's disease. Curr Alzheimer Res. 2007 Dec;4(5):550-2. doi: 10.2174/156720507783018217. PMID 18220520
- [Background] Tobinick EL. A critique of intradiscal administration for treatment of radiculopathy. Anesthesiology. 2008 Feb;108(2):334; author reply 335. doi: 10.1097/01.anes.0000300072.56020.10. No abstract available. PMID 18212586
- [Background] Tobinick E. Perispinal etanercept produces rapid improvement in primary progressive aphasia: identification of a novel, rapidly reversible TNF-mediated pathophysiologic mechanism. Medscape J Med. 2008 Jun 10;10(6):135. PMID 18679537
- [Background] Chainani-Wu N. Safety and anti-inflammatory activity of curcumin: a component of tumeric (Curcuma longa). J Altern Complement Med. 2003 Feb;9(1):161-8. doi: 10.1089/107555303321223035. PMID 12676044
- [Background] Pendurthi UR, Williams JT, Rao LV. Inhibition of tissue factor gene activation in cultured endothelial cells by curcumin. Suppression of activation of transcription factors Egr-1, AP-1, and NF-kappa B. Arterioscler Thromb Vasc Biol. 1997 Dec;17(12):3406-13. doi: 10.1161/01.atv.17.12.3406. PMID 9437186
- [Background] Antony S, Kuttan R, Kuttan G. Immunomodulatory activity of curcumin. Immunol Invest. 1999 Sep-Dec;28(5-6):291-303. doi: 10.3109/08820139909062263. PMID 10574627
- [Background] Jobin C, Bradham CA, Russo MP, Juma B, Narula AS, Brenner DA, Sartor RB. Curcumin blocks cytokine-mediated NF-kappa B activation and proinflammatory gene expression by inhibiting inhibitory factor I-kappa B kinase activity. J Immunol. 1999 Sep 15;163(6):3474-83. PMID 10477620
- [Background] Lim GP, Chu T, Yang F, Beech W, Frautschy SA, Cole GM. The curry spice curcumin reduces oxidative damage and amyloid pathology in an Alzheimer transgenic mouse. J Neurosci. 2001 Nov 1;21(21):8370-7. doi: 10.1523/JNEUROSCI.21-21-08370.2001. PMID 11606625
- [Background] Yang F, Lim GP, Begum AN, Ubeda OJ, Simmons MR, Ambegaokar SS, Chen PP, Kayed R, Glabe CG, Frautschy SA, Cole GM. Curcumin inhibits formation of amyloid beta oligomers and fibrils, binds plaques, and reduces amyloid in vivo. J Biol Chem. 2005 Feb 18;280(7):5892-901. doi: 10.1074/jbc.M404751200. Epub 2004 Dec 7. PMID 15590663
- [Background] Ueda H, Yamazaki C, Yamazaki M. Luteolin as an anti-inflammatory and anti-allergic constituent of Perilla frutescens. Biol Pharm Bull. 2002 Sep;25(9):1197-202. doi: 10.1248/bpb.25.1197. PMID 12230117
- [Background] Xagorari A, Papapetropoulos A, Mauromatis A, Economou M, Fotsis T, Roussos C. Luteolin inhibits an endotoxin-stimulated phosphorylation cascade and proinflammatory cytokine production in macrophages. J Pharmacol Exp Ther. 2001 Jan;296(1):181-7. PMID 11123379
- [Background] Rezai-Zadeh K, Douglas Shytle R, Bai Y, Tian J, Hou H, Mori T, Zeng J, Obregon D, Town T, Tan J. Flavonoid-mediated presenilin-1 phosphorylation reduces Alzheimer's disease beta-amyloid production. J Cell Mol Med. 2009 Mar;13(3):574-88. doi: 10.1111/j.1582-4934.2008.00344.x. Epub 2008 Apr 9. PMID 18410522
- [Background] Borchers AT, Sakai S, Henderson GL, Harkey MR, Keen CL, Stern JS, Terasawa K, Gershwin ME. Shosaiko-to and other Kampo (Japanese herbal) medicines: a review of their immunomodulatory activities. J Ethnopharmacol. 2000 Nov;73(1-2):1-13. doi: 10.1016/s0378-8741(00)00334-2. PMID 11025134
- [Background] Lo CJ, Chiu KC, Fu M, Lo R, Helton S. Fish oil decreases macrophage tumor necrosis factor gene transcription by altering the NF kappa B activity. J Surg Res. 1999 Apr;82(2):216-21. doi: 10.1006/jsre.1998.5524. PMID 10090832
- [Background] Lukiw WJ, Cui JG, Marcheselli VL, Bodker M, Botkjaer A, Gotlinger K, Serhan CN, Bazan NG. A role for docosahexaenoic acid-derived neuroprotectin D1 in neural cell survival and Alzheimer disease. J Clin Invest. 2005 Oct;115(10):2774-83. doi: 10.1172/JCI25420. PMID 16151530
- [Background] Yano M, Kishida E, Iwasaki M, Kojo S, Masuzawa Y. Docosahexaenoic acid and vitamin E can reduce human monocytic U937 cell apoptosis induced by tumor necrosis factor. J Nutr. 2000 May;130(5):1095-101. doi: 10.1093/jn/130.5.1095. PMID 10801904
- [Background] Calder PC. Immunomodulation by omega-3 fatty acids. Prostaglandins Leukot Essent Fatty Acids. 2007 Nov-Dec;77(5-6):327-35. doi: 10.1016/j.plefa.2007.10.015. Epub 2007 Nov 26. PMID 18032006
- [Background] Venkatraman JT, Chu WC. Effects of dietary omega-3 and omega-6 lipids and vitamin E on serum cytokines, lipid mediators and anti-DNA antibodies in a mouse model for rheumatoid arthritis. J Am Coll Nutr. 1999 Dec;18(6):602-13. doi: 10.1080/07315724.1999.10718895. PMID 10613412
- [Background] Caughey GE, Mantzioris E, Gibson RA, Cleland LG, James MJ. The effect on human tumor necrosis factor alpha and interleukin 1 beta production of diets enriched in n-3 fatty acids from vegetable oil or fish oil. Am J Clin Nutr. 1996 Jan;63(1):116-22. doi: 10.1093/ajcn/63.1.116. PMID 8604658
- [Background] James MJ, Gibson RA, Cleland LG. Dietary polyunsaturated fatty acids and inflammatory mediator production. Am J Clin Nutr. 2000 Jan;71(1 Suppl):343S-8S. doi: 10.1093/ajcn/71.1.343s. PMID 10617994
- [Background] Kotani S, Sakaguchi E, Warashina S, Matsukawa N, Ishikura Y, Kiso Y, Sakakibara M, Yoshimoto T, Guo J, Yamashima T. Dietary supplementation of arachidonic and docosahexaenoic acids improves cognitive dysfunction. Neurosci Res. 2006 Oct;56(2):159-64. doi: 10.1016/j.neures.2006.06.010. Epub 2006 Aug 14. PMID 16905216
- [Background] Freund-Levi Y, Eriksdotter-Jonhagen M, Cederholm T, Basun H, Faxen-Irving G, Garlind A, Vedin I, Vessby B, Wahlund LO, Palmblad J. Omega-3 fatty acid treatment in 174 patients with mild to moderate Alzheimer disease: OmegAD study: a randomized double-blind trial. Arch Neurol. 2006 Oct;63(10):1402-8. doi: 10.1001/archneur.63.10.1402. PMID 17030655
- [Background] Rosen WG, Terry RD, Fuld PA, Katzman R, Peck A. Pathological verification of ischemic score in differentiation of dementias. Ann Neurol. 1980 May;7(5):486-8. doi: 10.1002/ana.410070516. PMID 7396427